CLINICAL TRIAL: NCT02452320
Title: Prospective, Double Blind, Placebo Control, Study of Acetaminophen iv on Hospital Length of Stay in Morbidly Obese Individuals Undergoing Elective Laparoscopic Sleeve Gastrectomy
Brief Title: Prospective, Double Blind, Placebo Control, Bariatric IV Ace
Acronym: Bariatricace
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1503016056
Record Dates: First submitted 2015-05-04; First posted 2015-05-22 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Obesity
Keywords: bariatric; Post-operative nausea and vomiting; laparoscopic Sleeve gastrectomy; intravenous acetaminophen
MeSH Terms: conditions — Obesity; Vomiting | interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Subjects randomized into the control group will not receive study medication, they will receive a placebo administered at the same schedule as the active drug in the other arm.
  Interventions: Drug: Placebo
- Randomized (Active Comparator): Subjects randomized into the active treatment group will receive intravenous acetaminophen
  Interventions: Drug: intravenous acetaminophen

INTERVENTIONS:
Drug: intravenous acetaminophen — administration of 1000mg of intravenous acetaminophen or placebo every 6 hours for a total of 4 doses; first dose to be administered after induction of general anesthesia
  Other Names: Ofirmev
  Arms: Randomized
Drug: Placebo — Subjects randomized to placebo will receive every 6 hours for a total of 4 doses; first dose to be administered after induction of general anesthesia
  Other Names: Normal Saline
  Arms: Control

SUMMARY:
The purpose of this study is to determine if the administration of acetaminophen given intravenously (through an IV) beginning during surgery and then for 3 additional doses during the first 24 hours post-operatively will reduce the length of time subjects undergoing elective sleeve gastrectomy spend in the hospital following this operation. Additional questions that may be answered include whether administration of the study medication leads to improvement in pain control, a reduction in post-operative nausea and vomiting, and an overall improvement in quality of recovery.

DETAILED DESCRIPTION:
Morbid obesity is defined as a body mass index (BMI: weight [kg] / height [m]2) ≥ 40 or ≥ 35 if associated with comorbidities, and it is widely prevalent, nationally and globally. Overweight or obese individuals have increased morbidity and mortality. Among the many available treatment options, surgical management of obesity has been shown to be the most reliably effective in achieving sustained weight loss and improvements in glycemic, lipidemic, and blood pressure control, and improves five and ten year survival in contrast to matched controls who did not have surgery. Various surgical approaches have been used to provide long-term control of morbid obesity and its associated comorbidities, including laparoscopic sleeve gastrectomy.

During a sleeve gastrectomy the greater curvature of the stomach is separated from the lesser curvature and antrum, thereby eliminating ~85% of the total stomach, including the grehlin-producing portion of the stomach. A common complication of the procedure is postoperative nausea and vomiting (PONV), occurring in nearly 80% of patients undergoing the procedure. Risk factors for PONV include: female sex, history of PONV or motion sickness, nonsmoking, younger age, general vs. regional anesthesia, use of volatile anesthetics and nitrous oxide, administration of postoperative opioids, duration of anesthesia, and type of surgery (including cholecystectomy, laparoscopic, and gynecological). At the individual level, PONV adversely impacts both patient satisfaction and quality of life scores. At the systems level, PONV is associated with increased length of stay (LOS) in the post-anesthesia care unit and hospital, and can result in increased costs.

Both pharmacological and surgical approaches have been studied in an effort to reduce the incidence of PONV in sleeve gastrectomy patients. Omentopexy was unsuccessful, and pharmacologic prophylaxis with two [dexamethasone + odansetron; dexamethasone + granisetron; aprepitant + odansetron; or three (dexamethasone + odansetron + haloperidol; antiemetic agents was more effective than a single agent (odansetron or granisetron) alone in decreasing both nausea and vomiting. Even with triple therapy, just over 50% of patients were nauseous and 20% vomited within the first 36 hours following surgery, and hospital LOS was unaffected. Thus, there is a pressing need for improved control of PONV in sleeve gastrectomy patients.

Acetaminophen (N-(4-hydroxyphenyl)acetamide; paracetamol) is a mild analgesic whose main, but not sole, mechanism of action is thought to arise from inhibition of the cyclooxygenase pathway; the intravenous (iv) formulation (acetaminophen iv; ACP-iv) received US Food and Drug Administration (FDA) approval in November 2010 but has been available in Europe since 2002. It is approved by the FDA for the management of mild to moderate pain as a single agent and the management of moderate to severe pain with adjunctive opioid analgesics. Recently, two meta-analyses have evaluated the use of ACP-iv in the postoperative period for its efficacy in preventing postoperative pain [45] or reducing PONV [46]. In the study by De Oliveria et al., ACP-iv administration was found to significantly reduce postoperative pain, opioid consumption, and PONV. Similarly, the study by Apfel and colleagues indicated that iv-ACP, when administered prophylactically, reduced PONV as a consequence of improved pain control. With direct relevance to sleeve gastrectomy patients, a retrospective analysis of patients undergoing bariatric surgery (sleeve gastrectomy or laparoscopic Roux-en-Y gastric bypass) found that ACP-iv administration reduced opiate consumption and hospital LOS.

The investigators hypothesize that administration of ACP-iv in the perioperative period will reduce hospital LOS in sleeve gastrectomy subjects and will be associated with a reduction in hospital costs. The secondary hypothesis is that administration of ACP-iv will reduce PONV and improve subject satisfaction scores in the same subject population.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* BMI > 30
* Undergoing Elective Sleeve Gastrectomy
* Able to consent

Exclusion Criteria:

* Allergy/ Hypersensitive to acetaminophen or formulation incipients
* Allergy/Hypersensitive to aprepitant, ondasteron (serotonin type 3 receptor antagonists), dexamethasone
* Allergy to Propofol or formulation incipients (egg albumin, soy lecithin)
* Diagnosis or positive family history of malignant hyperthermia
* Abnormal LFTs (AST and ALT) >2x local upper limits of normal
* Renal impairment (creatinine clearance (CrCl) ≤ 30mL/min adjusted for obesity))
* Pregnancy
* Alcohol consumption > 3 drinks/day
* Requires awake intubation
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Goldstein, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
We will not be making IPD available

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 136 subjects were informed of and consented to participate. Due to unforeseen scheduling conflicts and canceled surgeries, we recruited more subjects in order to reach our 128 recruitment mark for statistical analysis.
  1 subject was not included in the analysis due to a prolonged hospitalization not related to the study.
Groups:
- Placebo: Subjects randomized into the control group will not receive study medication, they will receive a placebo administered at the same schedule as the active drug in the other arm.
  Placebo: Subjects randomized to placebo will receive every 6 hours for a total of 4 doses; first dose to be administered after induction of general anesthesia
- Acetaminophen IV: Subjects randomized into the active treatment group will receive intravenous acetaminophen
  intravenous acetaminophen: administration of 1000mg of intravenous acetaminophen or placebo every 6 hours for a total of 4 doses; first dose to be administered after induction of general anesthesia
Period: Overall Study
Arm/Group | Placebo | Acetaminophen IV
Started | 64 | 64
Completed | 64 | 63
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Acetaminophen IV | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (12.2) | 42.2 (12.2) | 40.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 45 | 92
  Male | 17 | 18 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: When added the breakdown of participants is equivalent to the overall number of participants
  Participants
    White: number analyzed (Participants) | 24 | 21 | 45
    White | 24 | 21 | 45
    Black or African American | 20 | 16 | 36
    More than one race | 7 | 13 | 20
    Unknown or Not Reported | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  United States | 64 | 63 | 127
Height (cm) [Mean (Standard Deviation); unit: cm] | 164.8 (10.8) | 165.5 (9.2) | 165.2 (10)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 130 (27.1) | 127.5 (25.4) | 128.8 (26.3)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 47.3 (7.9) | 46.6 (7.7) | 46.9 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery-15 Patient Survey
Description: Survey asking 15 questions with regard to how the patient is feeling scored on a scale from 0-10, with 0 being none of the time and 10 being all of the time. Possible scores range from 0-150, and scores with a higher value indicate a better outcome. Each subject was administered a baselineQoR-15 survey prior to surgery, and then one on postoperative days (POD) 1 and 2. If a subject was discharged prior to POD2, they were not given a QoR-15 survey that day.
Time Frame: Patients will be followed for the duration of hospital stay, expected average of 3 days.
Population: Subjects were administered a QoR-15 Survey pre-operatively as a baseline, and on post-operative days 1 and 2. Some subjects were discharged prior to the administration of the QoR-15 on post-operative day 2 and therefore there is no data for those subjects that we no longer in the hospital.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Acetaminophen IV
Number analyzed (Participants) | 64 | 63
units on a scale
  POD 1 | 107.2 (18.8) | 108.6 (20.9)
  POD 2 | 118.3 (17.3) | 117.1 (21.1)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen IV; Test type: Other; p = 0.59, t-test, 2 sided

2. Secondary Outcome: Length of Hospital Stay
Description: Monitoring the length of hospital stay after undergoing surgery
Time Frame: Participants will be followed for the duration of hospital stay, expected average of 3 days.
Population: Subjects LoS were recorded from time of PACU admission till time that Discharge Orders were completed.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Acetaminophen IV
Number analyzed (Participants) | 64 | 63
days | 1.96 [1.80 to 2.31] | 1.87 [1.66 to 2.06]

3. Secondary Outcome: Hospital Costs
Description: Accessing billing codes/hospital costs for each enrolled subject from the time they are admitted until they are discharged from the hospital.
Time Frame: Costs incurred during hospital stay, expected average of 3 days.
Population: Used the Hospital cost data for the subjects enrolled in both arms of the study for the duration of their hospitalization.
Measure: Median (Inter-Quartile Range); unit: Dollars (USD)
Arm/Group | Placebo | Acetaminophen IV
Number analyzed (Participants) | 64 | 63
Dollars (USD) | 12,977 [11,688 to 14,426] | 12,885 [11,376 to 15,226]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the time in which the subject was in the hospital. Our consent form allowed access to their electronic medical record while the subject was in the hospital. Adverse events were monitored while the subject was hospitalized, an average of 2-3 days. Once discharged from this hospitalization, the subjects were no longer followed.
Arm/Group | Placebo | Acetaminophen IV
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/64 | 1/63
Other Adverse Events (participants affected / at risk) | 0/64 | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=64) | Acetaminophen IV (N=63)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — One Subject (in the randomized arm) was admitted into the SICU post-op due to pulmonary complications unrelated to the study.

LIMITATIONS AND CAVEATS:
Limitations of this study: Did not follow subjects after discharge and therefore do not have any re-admission data (if applicable). Relatively small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No